CLINICAL TRIAL: NCT04201795
Title: Effects of the Pressure and Traction Technique on the Plantar Footprint and Balance Against a Placebo Laser: A Randomized Single Blind Trial
Brief Title: Effects of the Pressure and Traction Technique on the Plantar Footprint and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2111201814518
Record Dates: First submitted 2019-12-09; First posted 2019-12-17 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Foot; Manual Therapy
Keywords: fascia; myofascial; plantar fascia; postural balance; stabilometry; platform
MeSH Terms: interventions — Lasers; Pressure

STUDY DESIGN:
Intervention Model Description: two arms parallel ( intervention and control) will be randomized asigned to compare pressure and traction tecnique versus laser placebo
Who Masked: Participant
Masking Description: single blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pressure and traction (Experimental): pressure and traction durin 5 minutes will be applied in plantar fascia
  Interventions: Other: pressure and traction tecnique
- Laser (Sham Comparator): Applied during 5 minutes each plantar fascia of sham laser
  Interventions: Other: Laser

INTERVENTIONS:
Other: Laser — laser with no emision will applied
  Arms: Laser
Other: pressure and traction tecnique — pressure and traction in plantar fascia with hands will be applied
  Arms: pressure and traction

SUMMARY:
The aim of this clinical trial is to check the effects of manual pressure and traction technique on balance and plantar footprint variables comparing with Laser placebo.

DETAILED DESCRIPTION:
Forty healthy subjects wil be recruited for a simple blind study. Participants will be from 1 to 40 years old, not obese. Participants will be randomized into two groups. Experimental group performed a bilateral plantar fascia manual pressure and traction technique. Control group performed a laser placebo. The time duration (5 minutes), position, and therapist were the same for both treatments. The investigators will measure stabilometry variables and static footprint. The footprint variables will be divided in bilateral rear foot, bilateral midfoot, bilateral fore foot.

Measures. Stabilometry will be measured by displacement of the center of pressures in X and Y with eyes open and closed , center of pressure (COP) with eyes open and closed, COP area with eyes open and closed, COP antero-posterior (a-p) and medio-lateral (m-lat) directions with eyes open and closed, and COP speed. Two trials will be recorded for each condition and the order of the conditions will be randomized across subjects, eyes open and eyes closed. Foot plantar pressure and surface area of two static footprints will be measured during bipedal standing. Static plantar pressure will be evaluated by means of maximum pressure, medium pressure and surface area of each aspect of the foot (rearfoot, midfoot, and fore foot).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Must have no pain

Exclusion Criteria:

* Previous lower extremities surgery.
* History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.
* Leg-length discrepancy more than 1 cm
* Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
static footprint | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline
stabilometry variables eyes open | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform (27), participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes open
stabilometry variables eyes closed | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform (27), participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes closed

SECONDARY OUTCOMES:
static footprint after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline
stabilometry variables eyes open after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform (27), participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes open
stabilometry variables eyes after intervention | Through study completion, an average of 1 month
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform (27), participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. During all the examinations, the upper limbs were placed in a relaxed position along the body. The subjects were instructed to stand as still as possible for 30 s, with their eyes open, while concentrating on a point at eye level 2-m away or with their eyes closed

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez-Jimenez, Principal Investigator — Mayuben Clinic
Locations (1):
- Mayuben Clinic, San Sebastián de los Reyes, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajimsha MS, Binsu D, Chithra S. Effectiveness of myofascial release in the management of plantar heel pain: a randomized controlled trial. Foot (Edinb). 2014 Jun;24(2):66-71. doi: 10.1016/j.foot.2014.03.005. Epub 2014 Mar 21. PMID 24703512
- [Background] Ajimsha MS, Chithra S, Thulasyammal RP. Effectiveness of myofascial release in the management of lateral epicondylitis in computer professionals. Arch Phys Med Rehabil. 2012 Apr;93(4):604-9. doi: 10.1016/j.apmr.2011.10.012. Epub 2012 Jan 10. PMID 22236639
- [Background] Ichikawa K, Takei H, Usa H, Mitomo S, Ogawa D. Comparative analysis of ultrasound changes in the vastus lateralis muscle following myofascial release and thermotherapy: a pilot study. J Bodyw Mov Ther. 2015 Apr;19(2):327-36. doi: 10.1016/j.jbmt.2014.11.018. Epub 2014 Dec 23. PMID 25892389
- [Background] Hyland MR, Webber-Gaffney A, Cohen L, Lichtman PT. Randomized controlled trial of calcaneal taping, sham taping, and plantar fascia stretching for the short-term management of plantar heel pain. J Orthop Sports Phys Ther. 2006 Jun;36(6):364-71. doi: 10.2519/jospt.2006.2078. PMID 16776486
- [Background] Lee M, Kim M, Oh S, Choi YJ, Lee D, Lee SH, Yoon B. A self-determination theory-based self-myofascial release program in older adults with myofascial trigger points in the neck and back: A pilot study. Physiother Theory Pract. 2017 Sep;33(9):681-694. doi: 10.1080/09593985.2017.1345024. Epub 2017 Jul 17. PMID 28715296